CLINICAL TRIAL: NCT07149987
Title: Assessing the Role of 3D-Printed Surgical Guides in Enhancing Dental Implant Placement Precision and Patient Outcomes
Brief Title: Fully Guided Dental Implant Placement and Primary Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mosul (Other)
Responsible Party: Principal Investigator, Munib Abdullah Fathi, Assist.Prof.Dr. Munib Abdullah Fathi, University of Mosul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOM.Dent/25/1029; self-funded (Other: UOM-Oral and Maxillofacial surgery Department)
Record Dates: First submitted 2025-07-16; First posted 2025-09-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Dental Implant; Dental Implant Failure; Peri Implantitis; Cone Beam Computed Tomography
Keywords: 3D- implant surgical guide; C-Tech® implants; DICOM file
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Methods: randomized controlled clinical study included 30 patients with a total of 30 implants were placed and analyzed. All patients were randomly allocated into two groups: Test Group (Guided Surgery Group) and Control Group (Freehand Surgery Group). For all the patient in the study primary stability was assessed immediately after implant placement and secondary stability was assessed three months postoperatively. Postoperative pain was measured using the (VAS), immediately after surgery and one week later
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Guided Surgery Group) (Experimental): Test Group (Guided Surgery Group): Implants were placed using 3D-printed surgical guides
  Interventions: Procedure: All implant placements were performed exclusively in the maxillary region (upper jaw) to ensure a controlled comparison within the same anatomical area
- Control Group (Freehand Surgery Group) (No Intervention): Implants were placed freehand without guide assistance

INTERVENTIONS:
Procedure: All implant placements were performed exclusively in the maxillary region (upper jaw) to ensure a controlled comparison within the same anatomical area — All implant placements were performed exclusively in the maxillary region (upper jaw) to ensure a controlled comparison within the same anatomical area. The implants used in this study were C-Tech® implants (C-Tech Implant, Italy) with the following dimensions: Diameter: 3.8 mm Length: 11 mm . Cone-Beam Computed Tomography (CBCT): To assess bone quality, quantity, and anatomical structures . Digital Intraoral Scans Heron Scanner (USA) to obtain detailed gingival contours, occlusion, and existing teeth. The scan data was exported as an STL file for digital planning. Easy Check Implant Stability Measuring System is used for implant stability measurement, the tapping rod was gently placed in slight contact with the healing abutment, avoiding any axial or lateral pressure, and aligned within 0°-30° relative to the abutment's occlusal surface. If the angle exceeded 30°, the device issued an alert and prevented measurement, ensuring consistent alignment
  Arms: Test Group (Guided Surgery Group)

SUMMARY:
The precision of dental implant placement is vital for long-term implant success. The surgical guide is designed using advanced 3D imaging techniques allows for a highly accurate simulation of the ideal implant position, angulation, and depth based on the patient's unique anatomy. The aim of the study is to compare implant stability and postoperative pain between guided and freehand surgical implant placement. The research objective is to assess and compare the clinical outcomes of guided surgical implants placement versus conventional freehand implant placement, focusing on primary implant stability, secondary implant stability and postoperative pain. In alignment with this objective, the aim of this study is to compare the clinical outcomes: as implant primary and secondary stability and postoperative pain between guided surgical implant placement and conventional freehand surgical implant placement.

Hypothesis of the study This study hypothesized that guided implant surgery will result in superior implant stability outcome and reduced postoperative pain compared to the freehand technique High light of study. The use of advance technology (machines and software programs) to enhance implant survival and reduce surgical complications associated with implant placement. It is worth noting that, a fully guided implant placement provides flapless surgery and the implant positions were virtually planned based on anatomical and prosthetic considerations. The use of Easy Check Implant Stability Measuring System for measuring primary and secondary implant stability.

DETAILED DESCRIPTION:
Background: The precision of dental implant placement is vital for long-term implant success. The surgical guide is designed using advanced 3D imaging techniques allows for a highly accurate simulation of the ideal implant position, angulation, and depth based on the patient's unique anatomy. The aim of the study is to compare implant stability and postoperative pain between guided and freehand surgical implant placement.

Methods: randomized controlled clinical study included 30 patients with a total of 30 implants were placed and analyzed. All patients were randomly allocated into two groups: Test Group (Guided Surgery Group) and Control Group (Freehand Surgery Group). For all the patient in the study primary stability was assessed immediately after implant placement and secondary stability was assessed three months postoperatively. Postoperative pain was measured using the (VAS), immediately after surgery and one week later.

ELIGIBILITY:
The inclusion criteria for the study were:

1. Patients ≥18 years of age.
2. Presenting with maxillary tooth loss,
3. Tooth extraction at least 3 months before (delayed placement)
4. Adequate amount of bone volume to place the implant without bone augmentation (2 mm bone circumferentially around the implant).

The exclusion criteria for the study were: Patients were excluded from the study for the following reasons:

1. General contraindications to implant surgery;
2. Patients with history of chemo or radiotherapy;
3. Poor oral hygiene;
4. Pregnant or lactating women;
5. Uncontrolled diabetic patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
post operative pain | From placement of implant immediately and to the 2nd visit of treatment at one week
  Postoperative pain was measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain), immediately after surgery and one week later
primary stability improvement | For all the patient in the study primary stability was assessed immediately after implant placement
  For all the patient in the study primary stability was assessed postoperatively using ISQ. The Scale Implant Stability Quotient (ISQ) range between 1 to 100. The Interpretation of scores as follow:
  ISQ >70: High stability ISQ 60-69: Moderate stability ISQ <60: Low stability

SECONDARY OUTCOMES:
secondary stability outcome measure | For all the patient in the study, the secondary stability was assessed three months from implant placement
  the secondary stability was assessed using ISQ. The Scale Implant Stability Quotient (ISQ) range between 1 to 100. The Interpretation of scores as follow: ISQ >70: High stability ISQ 60-69: Moderate stability ISQ <60: Low stability

CONTACTS AND LOCATIONS:
Overall Officials: AbdAlhameed N. Aldabagh, AssistProfDr, Principal Investigator — Department of OMFS, College of Dentistry, University of Mosul, Nineveh, Iraq
Locations (1):
- University of Mosul/ College of Dentistry/ oral and Maxillofacial depart./Teaching dental Clinics unit/dental implant and laser unit, Mosul, Iraq

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared for this study due to ethical considerations and confidentiality regulations. The study protocol does not include plans for IPD sharing, in accordance with institutional and national data protection policies

REFERENCES:
- [Background] Marra R, Acocella A, Rispoli A, Sacco R, Ganz SD, Blasi A. Full-mouth rehabilitation with immediate loading of implants inserted with computer-guided flap-less surgery: a 3-year multicenter clinical evaluation with oral health impact profile. Implant Dent. 2013 Oct;22(5):444-52. doi: 10.1097/ID.0b013e31829f1f7f. PMID 24021974
- [Background] Barone A, Toti P, Piattelli A, Iezzi G, Derchi G, Covani U. Extraction socket healing in humans after ridge preservation techniques: comparison between flapless and flapped procedures in a randomized clinical trial. J Periodontol. 2014 Jan;85(1):14-23. doi: 10.1902/jop.2013.120711. Epub 2013 May 20. PMID 23688103
- [Background] Hultin M, Svensson KG, Trulsson M. Clinical advantages of computer-guided implant placement: a systematic review. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:124-35. doi: 10.1111/j.1600-0501.2012.02545.x. PMID 23062137
- [Background] Arisan V, Karabuda CZ, Ozdemir T. Implant surgery using bone- and mucosa-supported stereolithographic guides in totally edentulous jaws: surgical and post-operative outcomes of computer-aided vs. standard techniques. Clin Oral Implants Res. 2010 Sep;21(9):980-8. doi: 10.1111/j.1600-0501.2010.01957.x. Epub 2010 May 24. PMID 20497439
- [Background] Cassetta M, Bellardini M. How much does experience in guided implant surgery play a role in accuracy? A randomized controlled pilot study. Int J Oral Maxillofac Surg. 2017 Jul;46(7):922-930. doi: 10.1016/j.ijom.2017.03.010. Epub 2017 Mar 31. PMID 28366450
- [Background] Huang YC, Huang YC, Ding SJ. Primary stability of implant placement and loading related to dental implant materials and designs: A literature review. J Dent Sci. 2023 Oct;18(4):1467-1476. doi: 10.1016/j.jds.2023.06.010. Epub 2023 Jun 25. PMID 37799926
- [Background] Kim J, Park JY, Lee JY, Kim DM, Lee J, Jung UW, Lim YJ, Cha JK. Randomized controlled trial on the efficacy of a custom-made, fully guided implant system for flapless crestal sinus floor elevation: Accuracy and patient-reported outcomes. Clin Oral Implants Res. 2024 Dec;35(12):1531-1545. doi: 10.1111/clr.14341. Epub 2024 Aug 5. PMID 39101395
- [Background] Nagar P, Husain Z, Gupta U, Sheth M, Mishra R, Muthuraj HL. Comparative Study of Implant Placement Techniques and Their Effect on Long-Term Success of Implant-Supported Restorations. J Pharm Bioallied Sci. 2024 Dec;16(Suppl 4):S3500-S3502. doi: 10.4103/jpbs.jpbs_973_24. Epub 2024 Nov 13. PMID 39926875
- [Background] Rungcharassaeng K, Caruso JM, Kan JY, Schutyser F, Boumans T. Accuracy of computer-guided surgery: A comparison of operator experience. J Prosthet Dent. 2015 Sep;114(3):407-13. doi: 10.1016/j.prosdent.2015.04.004. Epub 2015 Jun 25. PMID 26119019
- [Background] Malo P, de Araujo Nobre M, Lopes A. The use of computer-guided flapless implant surgery and four implants placed in immediate function to support a fixed denture: preliminary results after a mean follow-up period of thirteen months. J Prosthet Dent. 2007 Jun;97(6 Suppl):S26-34. doi: 10.1016/S0022-3913(07)60005-5. Erratum In: J Prosthet Dent. 2008 Mar;99(3):167. PMID 17618930
- [Background] Di Giacomo GA, da Silva JV, da Silva AM, Paschoal GH, Cury PR, Szarf G. Accuracy and complications of computer-designed selective laser sintering surgical guides for flapless dental implant placement and immediate definitive prosthesis installation. J Periodontol. 2012 Apr;83(4):410-9. doi: 10.1902/jop.2011.110115. Epub 2011 Aug 5. PMID 21819249
- [Background] Moraschini V, Velloso G, Luz D, Barboza EP. Implant survival rates, marginal bone level changes, and complications in full-mouth rehabilitation with flapless computer-guided surgery: a systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2015 Jul;44(7):892-901. doi: 10.1016/j.ijom.2015.02.013. Epub 2015 Mar 17. PMID 25790741
- [Background] Ramakrishna R, Nayar S. Clinical assessment of primary stability of endosseous implants placed in the incisor region, using resonance frequency analysis methodology: an in vivo study. Indian J Dent Res. 2007 Oct-Dec;18(4):168-72. doi: 10.4103/0970-9290.35826. PMID 17938492
- [Background] Sul YT, Johansson CB, Jeong Y, Wennerberg A, Albrektsson T. Resonance frequency and removal torque analysis of implants with turned and anodized surface oxides. Clin Oral Implants Res. 2002 Jun;13(3):252-9. doi: 10.1034/j.1600-0501.2002.130304.x. PMID 12010155
- [Background] Javed F, Ahmed HB, Crespi R, Romanos GE. Role of primary stability for successful osseointegration of dental implants: Factors of influence and evaluation. Interv Med Appl Sci. 2013 Dec;5(4):162-7. doi: 10.1556/IMAS.5.2013.4.3. Epub 2013 Dec 20. PMID 24381734
- [Background] Bahrami R, Pourhajibagher M, Nikparto N, Bahador A. Robot-assisted dental implant surgery procedure: A literature review. J Dent Sci. 2024 Jul;19(3):1359-1368. doi: 10.1016/j.jds.2024.03.011. Epub 2024 Mar 19. PMID 39035318
- [Background] 20. Agha RA, Mathew G, Rashid R, Kerwan A, Al-Jabir A, Sohrabi C, Franchi T, Nicola M, Agha M, TITAN Group. Transparency In The reporting of Artificial INtelligence - the TITAN guideline. Premier Journal of Science 2025:10;100082
- [Background] Emery RW, Merritt SA, Lank K, Gibbs JD. Accuracy of Dynamic Navigation for Dental Implant Placement-Model-Based Evaluation. J Oral Implantol. 2016 Oct;42(5):399-405. doi: 10.1563/aaid-joi-D-16-00025. Epub 2016 Jun 6. PMID 27267658
- [Background] Chrcanovic BR, Kisch J, Albrektsson T, Wennerberg A. Factors Influencing Early Dental Implant Failures. J Dent Res. 2016 Aug;95(9):995-1002. doi: 10.1177/0022034516646098. Epub 2016 May 4. PMID 27146701
- [Background] Wahlberg RD, Stenport VF, Wennerberg A, Hjalmarsson L. A Multicenter Study of Factors Related to Early Implant Failures-Part 1: Implant Materials and Surgical Techniques. Clin Implant Dent Relat Res. 2025 Feb;27(1):e70015. doi: 10.1111/cid.70015. PMID 39976277
- [Background] Oh SH, Kim Y, Park JY, Jung YJ, Kim SK, Park SY. Comparison of fixed implant-supported prostheses, removable implant-supported prostheses, and complete dentures: patient satisfaction and oral health-related quality of life. Clin Oral Implants Res. 2016 Feb;27(2):e31-7. doi: 10.1111/clr.12514. Epub 2014 Oct 24. PMID 25346286
- [Background] Pjetursson BE, Bragger U, Lang NP, Zwahlen M. Comparison of survival and complication rates of tooth-supported fixed dental prostheses (FDPs) and implant-supported FDPs and single crowns (SCs). Clin Oral Implants Res. 2007 Jun;18 Suppl 3:97-113. doi: 10.1111/j.1600-0501.2007.01439.x. PMID 17594374
- [Background] Asghar AM, Sadaf D, Ahmad MZ, Jackson G, Bonsor SJ. Comparing clinical outcomes of immediate implant placement with early implant placement in healthy adult patients requiring single-tooth replacement in the aesthetic zone: a systematic review and meta-analysis of randomised controlled trials. Evid Based Dent. 2023 Jun;24(2):93. doi: 10.1038/s41432-023-00902-7. Epub 2023 Jun 5. PMID 37277486
- [Background] Kim Y, Oh TJ, Misch CE, Wang HL. Occlusal considerations in implant therapy: clinical guidelines with biomechanical rationale. Clin Oral Implants Res. 2005 Feb;16(1):26-35. doi: 10.1111/j.1600-0501.2004.01067.x. PMID 15642028
- [Background] Hopewell S, Chan AW, Collins GS, Hrobjartsson A, Moher D, Schulz KF, Tunn R, Aggarwal R, Berkwits M, Berlin JA, Bhandari N, Butcher NJ, Campbell MK, Chidebe RCW, Elbourne D, Farmer A, Fergusson DA, Golub RM, Goodman SN, Hoffmann TC, Ioannidis JPA, Kahan BC, Knowles RL, Lamb SE, Lewis S, Loder E, Offringa M, Ravaud P, Richards DP, Rockhold FW, Schriger DL, Siegried NL, Staniszewska S, Taylor RS, Thabane L, Torgerson D, Vohra S, White IR, Boutron I. CONSORT 2025 statement: Updated guideline for reporting randomised trials. PLoS Med. 2025 Apr 14;22(4):e1004587. doi: 10.1371/journal.pmed.1004587. eCollection 2025 Apr. PMID 40228477
- [Background] Chackartchi T, Romanos GE, Parkanyi L, Schwarz F, Sculean A. Reducing errors in guided implant surgery to optimize treatment outcomes. Periodontol 2000. 2022 Feb;88(1):64-72. doi: 10.1111/prd.12411. PMID 35103317
- [Background] Kumar Pandey A, Akkara F, Dhupar V. Efficacy of implant placement with surgical guides in the rehabilitation of the edentulous areas: An observational study and review of literature. Adv Oral Maxillofac Surg. 2022;8:100320
- [Background] Al Kabany MH. 3D-Printed Implant Sliding Guide: A New Dental Implant Surgical Guide. Int J Oral Maxillofac Implants. 2023 Oct 17;38(5):874-884. doi: 10.11607/jomi.10271. PMID 37847829
- [Background] Yeung M, Abdulmajeed A, Carrico CK, Deeb GR, Bencharit S. Accuracy and precision of 3D-printed implant surgical guides with different implant systems: An in vitro study. J Prosthet Dent. 2020 Jun;123(6):821-828. doi: 10.1016/j.prosdent.2019.05.027. Epub 2019 Oct 23. PMID 31653399
- [Background] Huang L, Liu L, Yang S, Khadka P, Zhang S. Evaluation of the accuracy of implant placement by using implant positional guide versus freehand: a prospective clinical study. Int J Implant Dent. 2023 Dec 1;9(1):45. doi: 10.1186/s40729-023-00512-z. PMID 38036932
- [Background] Corbella S, Morandi B, Calciolari E, Alberti A, Francetti L, Donos N. The influence of implant position and of prosthetic characteristics on the occurrence of peri-implantitis: a retrospective study on periapical radiographs. Clin Oral Investig. 2023 Dec;27(12):7261-7271. doi: 10.1007/s00784-023-05303-9. Epub 2023 Nov 1. PMID 37910236
- [Background] Chen ST, Buser D, Sculean A, Belser UC. Complications and treatment errors in implant positioning in the aesthetic zone: Diagnosis and possible solutions. Periodontol 2000. 2023 Jun;92(1):220-234. doi: 10.1111/prd.12474. Epub 2023 Jan 22. PMID 36683018
- [Background] Greenberg AM. Digital technologies for dental implant treatment planning and guided surgery. Oral Maxillofac Surg Clin North Am. 2015 May;27(2):319-40. doi: 10.1016/j.coms.2015.01.010. PMID 25951962
- [Background] Buser D, Martin W, Belser UC. Optimizing esthetics for implant restorations in the anterior maxilla: anatomic and surgical considerations. Int J Oral Maxillofac Implants. 2004;19 Suppl:43-61. PMID 15635945
- [Background] Esposito M, Hirsch JM, Lekholm U, Thomsen P. Biological factors contributing to failures of osseointegrated oral implants. (II). Etiopathogenesis. Eur J Oral Sci. 1998 Jun;106(3):721-64. doi: 10.1046/j.0909-8836..t01-6-.x. PMID 9672097
- [Background] Branemark PI, Hansson BO, Adell R, Breine U, Lindstrom J, Hallen O, Ohman A. Osseointegrated implants in the treatment of the edentulous jaw. Experience from a 10-year period. Scand J Plast Reconstr Surg Suppl. 1977;16:1-132. No abstract available. PMID 356184
- See also: The official website of C-Tech Implant (www.c-tech-implant.com) provides comprehensive and up-to-date information on the company's range of dental implant systems and accessories. — https://www.c-tech-implant.com/wp-content/uploads/download-prodotti/BL_surgical_protocol.pdf

DOCUMENTS (2):
  • Study Protocol (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT07149987/Prot_000.pdf
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT07149987/ICF_001.pdf